CLINICAL TRIAL: NCT06188546
Title: Administration of Propofol for Prophylaxis of Intrathecal Morphine Induced Pruritus in Caesarean Section
Brief Title: Propofol for Prophylaxis of Morphine Induced Pruritis in Caesarean Section
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sohila Khaled Mohamed Hassan, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: propofol for pruritis
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pruritus Caused by Drug
Keywords: morphine induced pruritus
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 0 (Placebo Comparator): Will receive no drugs for pruritis prophylaxis
  Interventions: Drug: Propofol
- Group 1 (Active Comparator): Will receive 1ml of propofol 10 mg/ml
  Interventions: Drug: Propofol
- Group 2 (Active Comparator): Will receive 2 ml of propofol 10mg/ml
  Interventions: Drug: Propofol
- Group 3 (Active Comparator): Will receive 3 ml of propofol 10mg/ml
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — trying different dosages of propofol 10mg/ml IV to determine the prophylactic dose for morphine induced pruritis

SUMMARY:
the goal of this randomized clinical trial is to find the optimum sub hypnotic dose of iv propofol that prevents the incidence of itching induced from intrathecal morphine used in spinal anesthesia in caesarean section operation. the main questions it aim to answer are the number of patients complained of pruritus in the first 24 hours post operative period and the severity of the pruritus. participants will be divided into 4 groups. 1st group receives 0 mg of propofol , 2nd receives 10 mg , 3rd receives 20 mg and the 4th receives 30 mg.

ELIGIBILITY:
Inclusion Criteria:

1. The study is scheduled for women undergoing elective caesarean section under spinal anesthesia.
2. The subject is ≥ 20 years and ≤ 40 years.
3. No obvious abnormalities in preoperative ECG, blood routine, electrolytes, and other tests.
4. ASA class 1-2.

Exclusion Criteria:

* Patients who had a known allergy to propofol, morphine, or bupivacaine.
* Those with preexisting pruritus caused by pregnancy, a coexisting skin disorder, or other pruritogenic systemic diseases.
* Patients with a contraindication to spinal anaesthesia
* Failed block
* Need of extra sedation intra-operative
* Positive history for asthma or COPD.
* Patient refusal

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
number of participants complained of pruritus in the first 24hr post operative period | first 24 hours post operative period

CONTACTS AND LOCATIONS:
Overall Officials: Zein Zarea, MD, Study Chair — Assiut University; Diab Fuad Hetta, MD, Study Director — South Egypt's cancer institute; Rania Mohamed Abdelemam, MD, Study Director — South Egypt's cancer institute

IPD SHARING:
Plan to Share IPD: No